CLINICAL TRIAL: NCT04197739
Title: Safety and Efficacy of Fixed-low-dose Amikacin for Urinary Tract Infection on the Elderly Patient
Brief Title: Fixed-dose Amikacin for Elderly UTI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-0619-19
Record Dates: First submitted 2019-12-08; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Urinary Tract Infections; Elderly Infection
Keywords: Urinary Tract Infections; Aminoglycosides; Amikacin; Elderly
MeSH Terms: conditions — Urinary Tract Infections | interventions — Amikacin

STUDY DESIGN:
Intervention Model Description: A randomized prospective, open label, non-inferiority trial
  Study participants will be 65 years or older, who were admitted to the medical ward due to a UTI will be assigned to one of the following study arms:
  1. Intervention arm: in which patients will receive a fixed dose of amikacin, 500 mg, once a day.
  2. Comparator arm: in which patients will receive a weight adjusted dose of amikacin (15 mg/kg adjusted body weight) and continue in adjusted intervals according plasma concentrations, using the Barnes Jewish Hospital nomogram.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed dose (Experimental): patients will receive a fixed, single daily dose of amikacin, 500 mg, a day.
  Interventions: Drug: Amikacin
- Adjusted body weight dose (Active Comparator): patients will receive a weight adjusted dose of amikacin (15 mg/kg adjusted body weight) and continue in adjusted intervals according to the Barnes Jewish Hospital nomogram.
  Interventions: Drug: Amikacin

INTERVENTIONS:
Drug: Amikacin — Patients in the intervention arm will receive a fixed, single daily dose of amikacin, 500 mg, a day.
  Patients in the Comparator arm will receive a weight adjusted loading dose of amikacin (15 mg/kg adjusted body weight) and continue in adjusted intervals according to the Barnes Jewish Hospital nomogram

SUMMARY:
Aminoglycosides are broad-spectrum antibiotics, effective against gram-negative bacteria. Aminoglycosides urine concentration exceeds that of the plasma by up to a hundred. Their efficacy is dependent on their level above minimal inhibitory concentration (MIC); however high levels are associate with nephrotoxicity. Therefore aminoglycosides have a narrow therapeutic rang. The correlation between administrated dose and blood drug levels is hard to predict. Amikacin is a highly effective aminoglycoside, highly effective against extended spectrum beta lactamase (ESBL) bacteria.

Older patients suffer from more urinary tract infection (UTIs), and have a higher frequency of infection with resistant bacteria, mainly among frail nursing home residents.

Our goal is to prove that fixed low dose amikacin in the elderly patient in non-inferior to weight-adjusted treatment.

Study design:

A randomized prospective, open label, non-inferiority trial

Study participants will be 65 years or older, who were admitted to the medical ward due to a UTI will be assigned to one of the following study arms:

1. Intervention arm: in which patients will receive a fixed dose of amikacin, 500 mg, once a day.
2. Comparator arm: in which patients will receive a weight adjusted dose of amikacin (15 mg/kg adjusted body weight) and continue in adjusted intervals according plasma concentrations, using the Barnes Jewish Hospital nomogram.

All participants will be followed up with:

1. Amikacin blood levels 6-14 hours following first administration, used for dose adjustment according to the nomogram. Peak amikacin blood levels, 30- 60 minutes following first or second administration.
2. Urine analysis and culture upon admission to the emergency department (ER). In patients with indwelling urinary catheters, cultures will be taken following replacement with a new catheter.
3. Broad serum biochemistry, complete blood count, C-reactive protein and blood cultures will be taken upon admission to the ER, two days after recruitment and at least once every three days following that, as long as the patient is receiving amikacin.

Duration of amikacin treatment will be according to the attending physician's clinical judgment; however, it will not be shorter than 72 hours since first dose. Total duration of amikacin treatment will not exceed 10 days. Total treatment for UTI will not fall short of seven days of antibiotics (either amikacin or any suitable alterative according to blood and/or urine cultures).

DETAILED DESCRIPTION:
Study protocol: Safety and efficacy of fixed-low-dose amikacin for urinary tract infection on the elderly patient.

Aminoglycosides are broad-spectrum, bactericidal antibiotics, effective against gram-negative bacteria. Of this group, gentamicin and amikacin are frequently used in our center (Rabin Medical Center, Beilinson campus). Amikacin, a semi-synthetic aminoglycoside, is highly effective against extended spectrum beta lactamase (ESBL) bacteria, and is the most effective against aminoglycoside modifying enzymes resistance.

Aminoglycosides are water soluble and mainly eliminated through the kidney. Their urine concentration exceeds that of the plasma up to a hundred. Aminoglycosides have a narrow therapeutic range, and the correlation between administrated dose and blood drug levels is hard to predict. Aminoglycosides' efficacy is dependent on their level above minimal inhibitory concentration (MIC). Common clinical practice regarding amikacin today is to administer a weight adjusted first dose, later measuring the blood drug level and adjusting following doses according to a nomogram (such as the Barnes Jewish Hospital nomogram). The evidence base behind the usage of the nomogram is lacking at best.

Our main concern with aminoglycosides is nephrotoxicity; amikacin was found to be less nephrotoxic than gentamycin. The nephrotoxic effect is dependent on the cumulative dose, and is documented mainly in association with high doses and long treatment courses.

On the one hand, elderly patients suffer from more urinary tract infection (UTIs), and have a higher frequency of infection with resistant bacteria. This latter problem is on the rise especially among frail and elderly nursing home residents. On the other hand, elderly patients are more prone to nephrotoxicity from aminoglycosides, due to the age-related decrease in glomerular filtration rate (GFR), polypharmacy and comorbidities. There is a true and vast lack of clinical trials regarding amikacin use in elderly patients, especially those aged 75 years or older.

Our goal is to prove that fixed low dose amikacin in the elderly patient in non-inferior to weight-adjusted treatment.

The investigators hypothesize that the use of fixed dose, 500 mg of amikacin, in the elderly will cause less nephrotoxicity and less dose-adjusting, with no more clinical failures.

Study participants will be 65 years or older, who were admitted to the medical ward due to a UTI.

Study design:

This is a prospective, open label, non-inferiority trial, in which consenting patients will be randomly assigned to one of the following study arms:

1. Intervention arm: in which patients will receive a fixed, single daily dose of amikacin, 500 mg, a day.
2. Comparator arm: in which patients will receive a weight adjusted loading dose of amikacin (15 mg/kg adjusted body weight) and continue in adjusted intervals according to the Barnes Jewish Hospital nomogram.

All participants will be followed up with:

1. Amikacin blood levels 6-14 hours following first administration after recruitment, used for dose adjustment according to the nomogram. Peak amikacin blood levels, 30- 60 minutes following first or second administration.
2. Urine analysis and urine culture upon admission to the emergency department (ER) (prior to recruitment). In patients with indwelling urinary catheters, cultures will be taken following replacement with a new catheter.
3. Broad serum biochemistry, complete blood count, C-reactive protein and blood cultures will be taken upon admission to the ER, two days after recruitment and at least once every three days following that, as long as the patient is receiving amikacin.

If in the intervention arm, serum amikacin levels will be found to be higher than that recommended for single daily dose (meaning toxic levels), the dosing intervals will also be adjusted according to the Barnes Jewish Hospital nomogram.

Duration of amikacin treatment will be according to the attending physician's clinical judgment; however, it will not be shorter than 72 hours since first dose. Total duration of amikacin treatment will not exceed 10 days. Total treatment for UTI will not fall short of seven days of antibiotics (either amikacin or any suitable alterative according to blood and/or urine cultures).

In both study arms, dosage or time interval adjustments and antibiotic type changes will be done only in the presence of lacking clinical improvement or according to blood and/or urine cultures.

No. of patients to be recruited: 200. Ages: 65 years or older. Sex: male or female.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of UTI according to: pyuria, along with a new complaint of dysuria, urgency or frequency of urination, or lower abdominal pain or discomfort; AND one of the following: systemic fever, flank pain, tenderness over the costo-vertebral angle, rigors and chills, vomiting.
2. Patients with moderate to severe cognitive impairment, who are unable to give reliable anamnesis, or those with permanent indwelling urinary catheter for 24 hours or more, will be considered as suffering from UTI is they present with systemic fever, pyuria and the lack of a more probable infectious cause.
3. Patients who can give informed consent or those with a legal guardian who can consent on their behalf.
4. Patients who received a single dose of any antimicrobial drug prior to recruitment, including amikacin.

   -

Exclusion Criteria:

1. Creatinine clearance < 40 mL/sec according to the Cockcroft-Gault equation
2. A known sensitivity to aminoglycosides
3. A known neuromuscular pathology (including myasthenia gravis).
4. Polycystic kidney disease
5. A urine or blood culture positive for amikacin resistant bacteria in the 30 days prior to recruitment.
6. Clinical suspicion of prostatitis, epididymitis or orchitis.
7. Hemodynamical instability (mean arterial pressure of 65 mmHg or under).
8. More than one dose of antimicrobial treatment that is adequate for classical UTI bacteria, unless a bacterial culture shows resistance to said treatment.
9. Immunosuppressed patients; steroidal treatment will be allowed.

   -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Composite clinical failure | 30 days
  A composite outcome of: clinical failure on day 5, all cause mortality on day 30, 30 days recurrent UTI.

SECONDARY OUTCOMES:
Rate of time-interval changes between amikacin doses | 5 days
  Incidence of time-interval changes between amikacin doses according to the Barnes Jewish Hospital nomogram.
Rates of antimicrobial drug change | 7-14 days
  Rates of antimicrobial drug change due to any cause
Clinical failure at day 5 | 5 days
  Persistent fever after 72 hours of treatment
Safety: acute kidney injury | 7-14 days
  Acute kidney injury according to the RIFLE criteria
Vestibular toxicity | 7-14 days
  New complaints of dizziness or giddiness